CLINICAL TRIAL: NCT05555199
Title: Injection of 99mTc-nanocolloid and ICG to Identify, Retrieve and Qualify Tumor Draining Lymph Nodes in Early-stage Lung Cancer
Brief Title: Injection of 99mTc-nanocolloid and ICG to Identify, Retrieve and Qualify TDLN in Early-stage NSCLC
Acronym: INITIATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Philips Healthcare (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 113036; NL81008.000.22 (Other: CCMO)
Record Dates: First submitted 2022-05-31; First posted 2022-09-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-04

CONDITIONS: Early-stage Lung Cancer
Keywords: Sentinel Lymph Node procedure; 99mTc-nanocolloid; ICG; SPECT/CT-imaging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, non-randomized, interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): One interventional arm that will undergo all interventional procedures (when applicable).
  Interventions: Radiation: 99mTc-nanocolloid; Drug: ICG

INTERVENTIONS:
Radiation: 99mTc-nanocolloid — Injection of 99mTc-nanocolloid when lung cancer is diagnosed during a navigation bronchoscopy, followed by one or two SPECT/CT-scans.
  Other Names: Elective navigation bronchoscopy; SLN procedure
Drug: ICG — If patient undergoes surgery to treat the lung cancer, ICG will be injected and retrieved fluorescent lymph nodes will undergo additional pathological assessment.
  Other Names: Elective lung surgery; SLN procedure

SUMMARY:
The patient wil receive intra- or peritumoral injections of 99mTc-nanocolloid if malignancy is found during a navigation bronchoscopy. A SPECT/CT-scan will be made to image injections sites and sentinel lymph nodes (SLN). If surgery takes place to treat the lung cancer, ICG will be injected and fluorescent lymph nodes will be extensively assessed by a pathologist.

DETAILED DESCRIPTION:
When malignancy is found during navigation bronchoscopy, study participants will receive intra- or peritumoral injections of 99mTc-nanocolloid. Following, up to 2 SPECT/CT-scans will be made to assess drainage of the injected tracer to the lymph nodes.

If patients undergo resection of the lung lesion, ICG will be injected. The involved lung tissue will be removed, followed by routine complete lymph node dissection. The fluorescent lymph nodes will be more extensively evaluated by the pathologist.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3;
* Lung lesion between 1 and 5 cm;
* Imaging-based disease free lymph nodes (N0);
* Patient is deemed a candidate for definitive lung tissue resection by a thoracic surgeon.

Exclusion Criteria:

* Pregnancy;
* Inability to consent;
* Known or suspected allergy to 99mTc-nanocolloid or ICG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of SLN procedure | During the study intervention
  This is a qualitative outcome measurement that will be assessed by the involved physicians based on the ability to inject 99mTc-nanocolloid and ICG, and the ability to detect the tumor draining lymph nodes based on their drainage patterns.

SECONDARY OUTCOMES:
Successfulness of injection method (intra- or peritumoral) | During the first intervention
Number of SLN found by SPECT/CT-imaging | On the day of the first intervention
Number of SLN found by ICG | On the day of the second intervention
Number of metastasis found by additional pathology | Up to two weeks after the second intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erik HF van der Heijden, Dr., Principal Investigator — Radboud University Medical Center; Desi KM ter Woerds, MSc., Study Director — Radboud University Medical Center; Roel LJ Verhoeven, Dr., Study Director — Radboud University Medical Center; Erik HJ Aartnzen, Dr., Study Director — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
(Pseudonymized) metadata will be stored for reuse and/or verification.
Supporting Information: Study Protocol
Time Frame: Data will be accessible for an unknown time after publication of the results.
Access Criteria: Under reasonable request.

REFERENCES:
- [Background] Sun WYL, Dang JT, Modasi A, Nasralla A, Switzer NJ, Birch D, Turner SR, Karmali S. Diagnostic accuracy of sentinel lymph node biopsy using indocyanine green in lung cancer: a systematic review and meta-analysis. Gen Thorac Cardiovasc Surg. 2020 Sep;68(9):905-913. doi: 10.1007/s11748-020-01400-8. Epub 2020 Jun 16. PMID 32557077
- [Background] Taghizadeh Kermani A, Bagheri R, Tehranian S, Shojaee P, Sadeghi R, N Krag D. Accuracy of sentinel node biopsy in the staging of non-small cell lung carcinomas: systematic review and meta-analysis of the literature. Lung Cancer. 2013 Apr;80(1):5-14. doi: 10.1016/j.lungcan.2013.01.001. Epub 2013 Jan 23. PMID 23352034
- [Background] Gilmore DM, Khullar OV, Colson YL. Developing intrathoracic sentinel lymph node mapping with near-infrared fluorescent imaging in non-small cell lung cancer. J Thorac Cardiovasc Surg. 2012 Sep;144(3):S80-4. doi: 10.1016/j.jtcvs.2012.05.072. Epub 2012 Jun 20. PMID 22726707
- [Background] Rena O, Boldorini R, Papalia E, Turello D, Massera F, Davoli F, Roncon A, Baietto G, Casadio C. Metastasis to subsegmental and segmental lymph nodes in patients resected for non-small cell lung cancer: prognostic impact. Ann Thorac Surg. 2014 Mar;97(3):987-92. doi: 10.1016/j.athoracsur.2013.11.051. Epub 2014 Jan 28. PMID 24480258